CLINICAL TRIAL: NCT01631578
Title: Phase 1 Study of the Impact of Injecting an Autologous Somatic Mitochondrial Concentrate Into Poor Quality Ova.
Brief Title: Improving the Reproductive Outcome of Poor Quality Ova by Injection of Autologous Somatic Mitochondria
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PI moved from medical center
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 252399- HMO-CTIL
Record Dates: First submitted 2012-05-24; First posted 2012-06-29 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Low Ovarian Reserve; Poor Quality Oocytes
Keywords: mitochondrial injection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Injection of mitochondrial concentrate (Experimental): A small volume of mitochondrial concentrate will be injected together with the spermatozoon during ICSI.
  Interventions: Procedure: Injection of an autologous mitochondria to the oocyte.
- Control (Active Comparator): ICSI will be performed conventionally.
  Interventions: Procedure: Injection of an autologous mitochondria to the oocyte.

INTERVENTIONS:
Procedure: Injection of an autologous mitochondria to the oocyte. — In the experimental group an autologous mitochondrial concentrate will be injected together with the sperm during ICSI. In the control group conventional ICSI will be performed.

SUMMARY:
A prospective randomized controlled trial (RCT) to determine the effect of injecting an autologous somatic mitochondria concentrate, together with the spermatozoon during ICSI, into oocytes of older and or poor prognosis in vitro fertilization (IVF) patients.

DETAILED DESCRIPTION:
Maternal age at first delivery constantly rises in developed countries. Oocyte quality decreases with advanced age, thus the rate of age-related infertility continuously increases. Presently oocyte donation is the only prompt solution for this widespread problem. Deterioration of mitochondrial function was suggested as one of the explanations for the age-related deterioration of oocyte quality. The supplementation of the ageing oocyte with autologous mitochondria from dividing somatic cells can be a possible solution for energetic enrichment, without introducing foreign mtDNA.

We established a non-hazardous clinical grade system to prepare functional autologous mitochondria concentrate from the granulosa cells aspirated during oocyte pick up. The mitochondrial preparation was examined and found to be non-toxic. The activity of the respiratory chain was constant and unaffected by age or ovarian response. Moreover, the mtDNA in the mitochondrial preparation was found to be intact in all samples examined, including those from older and low responding patients.

ELIGIBILITY:
Inclusion Criteria:

* Adequate sperm source and uterine cavity. And one or more of the following:
* Age > 40
* 3 unsuccessful IVF cycles or
* > 75% of embryos in previous cycles with > 20-50% fragments or
* < 50% fertilization rate in previous cycles

Exclusion Criteria:

* Inadequate sperm source. Inadequate uterine cavity.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Oocyte fertilization rate | one day
  Fertilization rate is assessed the day following oocyte retrieval.
The rate pace and quality of the early embryonic development | up to 6 days
  The rate (the proportion of fertilized oocytes developing into embryos), pace of cleavage, and quality (morphological) of the early embryonic development will be assessed during the next 1-6 days (case specific).

SECONDARY OUTCOMES:
Clinical pregnancy | within 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Yoel Shufaro, MD PhD, Principal Investigator — Hadassah
Locations (1):
- Hadassah University Hospital, Jerusalem, Israel